CLINICAL TRIAL: NCT05641090
Title: Effects of Nordic Walking in Water on Cerebrovascular Function and Cognitive Impairment in Elderly With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Prof. Dr.Daroonwan Suksom, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC-8
Record Dates: First submitted 2022-07-14; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Elderly With Type 2 Diabetes
Keywords: Type 2 Diabetes mellitus; Cerebrovascular function; Cognitive impairment; Nordic walking in water; Physical fitness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction | interventions — Nordic Walking; Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic walking in water (Experimental): The groups trained Nordic walking in water
  Interventions: Other: Nordic walking in water; Other: No exercise intervention
- No exercise intervention (No Intervention): The groups did not receive exercise

INTERVENTIONS:
Other: Nordic walking in water — Nordic walking in water will be based on nordic walking in water at temperature 34◦C. Nordic walking in water will be conducted at moderate intensity (40-60% heart rate reserve). The program was exercised 60 minutes include warm-up and cool down. At first 6 weeks, The exercise intensity was 40-50% heart rate reserve and it will be increased 50-60% heart rate reserve. The training program will be performed 3 times per week for 12 weeks.
  Arms: Nordic walking in water
Other: No exercise intervention — This group wasn't receive intervention program. The participants in this group will do following a physician who treat them. They can exercise according to the physician recommend.
  Arms: Nordic walking in water

SUMMARY:
Nordic walking in water would more advantage than normal daily life in cerebrovascular function and cognitive function in elderly with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included type 2 diabetes (as defined by the American Diabetes Association), a baseline glycosylated hemoglobin (HbA1c) value of 7-9%, and no previous exercise training in the past 6 months. All participants were free from diabetic nephropathy, diabetic retinopathy, severe diabetic neurophathy, severe cardiovascular and cerebrovascular diseases.
* Participants had Montreal Cognitive Assessment - Thai (MoCa-T) scores between 18 24 points.
* Participants had time up & go test between 8 - 15 seconds

Exclusion Criteria:

* Participants were excluded if they dropped out or completed less than 80% of the training schedule

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-04-05 (Estimated)

PRIMARY OUTCOMES:
General physiological data | Change from baseline systolic blood pressure, diastolic blood pressure, and mean arterial pressure at 12 weeks.
  1.Blood pressure in mmHg will be measured with automated blood pressure device (CARESCAPE V100, GE Dinamap).
Heart rate | Change from baseline heart rate at 12 weeks.
  Heart rate in beats per minute will be measured with automated blood pressure device (CARESCAPE V100, GE Dinamap).
ฺBody fat | Change from baseline body fat at 12 weeks.
  Body fat in percent will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcare).
Muscle mass and Weight | Change from baseline muscle mass and weight at 12 weeks.
  Muscle mass and weight in kilograms will be measured with dual energy x-ray absorptiometry (Prodigy-Pro, GE healthcare).
Arterial stiffness | Change from baseline brachial-ankle pulse wave velocity at 12 weeks.
  Arterial stiffness will be measured with brachial-ankle pulse wave velocity in centimeter per second (VP-1000 plus, omrom Healthcare).
Macro vascular function | Change from baseline brachial artery flow-mediated dilatation at 12 weeks.
  Macro vascular function will be measured by brachial artery flow-mediated dilatation in percent with ultrasonography equipment (EPIQ 5G, Phillips).
Cerebral blood flow | Change from baseline cerebral blood flow at 12 weeks.
  Cerebral blood flow in centimeter per second will be measured with ultrasonography equipment (EPIQ 5G, Phillips).
Cerebrovascular conductance index | Change from baseline cerebrovascular conductance index at 12 weeks.
  Cerebrovascular conductance index in cm/sec/mmHg will be measured with ultrasonography equipment (EPIQ 5G, Phillips).
Cerebrovascular reactivity index | Change from baseline cerebrovascular reactivity index at 12 weeks.
  Cerebrovascular reactivity index in %cm/sec/mmHg will be measured with ultrasonography equipment (EPIQ 5G, Phillips).
Arterial compliance | Change from baseline Arterial compliance at 12 weeks.
  Arterial compliance in units will be measure by carotid diameter during systolic and diastolic with ultrasonography equipment (EPIQ 5G, Phillips) and systemic blood pressure with (VP-1000 plus, omrom Healthcare).
Pulsatility index | Change from baseline Pulsatility index at 12 weeks.
  Pulsatility index in units will be measure with ultrasonography equipment (EPIQ 5G, Phillips).
Montreal Cognitive Assessment | Change from baseline Montreal Cognitive Assessment at 12 weeks.
  Montreal Cognitive Assessment in score (0 - 30 scores) cut off below 25 scores that indicate impairment cognitive function.
Mini-Mental State Examination | Change from baseline Mini-Mental State Examination at 12 weeks.
  Mini-Mental State Examination in scores (0 - 30 scores) cut off below 25 scores that indicate impairment cognitive function.
Trail Making Test-B and Stroop test | Change from baseline Trail Making Test-B and Stroop test at 12 weeks.
  Trail Making Test-B in second cut off below 101 seconds that indicate dementia. Stroop test in second will be measured with EncephalApp Stroop test.

SECONDARY OUTCOMES:
Waist circumference | Change from baseline waist circumference at 12 weeks
  Waist circumference in centimeters will be measure by waist tape
Flexibility testing | Change from baseline Chair sit & reach and Back scratch at 12 weeks.
  Flexibility testing will be measure by Chair sit & reach protocol and Back scratch in centimeters.
Muscle strength testing | Change from baseline arm-curl and chair stand at 12 weeks.
  Muscle strength testing will be measured by arm-curl test and chair stand test in repetitions in 30 seconds.
Balance testing | Change from baseline time up and go at 12 weeks.
  Balance testing will be measured by time up and go testing in seconds.
Cardiopulmonary fitness | Change from baseline 2-minutes step at 12 weeks.
  Cardiopulmonary fitness will be measure by 2-minutes step test in repetitions.
Cardiopulmonary fitness | Change from baseline 6-minutes walk at 12 weeks.
  Cardiopulmonary fitness will be measure by 6-minutes walk test in meters.
Fasting blood sugar | Change from baseline fasting blood sugar at 12 weeks.
  Fasting blood sugar in mg/dl will be measure with enzymatic assay using hexokinase reaction.
Glycosylated hemoglobin | Change from baseline Glycosylated hemoglobin at 12 weeks.
  Glycosylated hemoglobin in percent will be measure with enzymatic assay using hexokinase reaction.
Homeostasis Model Assessment of insulin resistance | Change from baseline Homeostasis Model Assessment of insulin resistance at 12 weeks.
  Homeostasis Model Assessment of insulin resistance in units will be calculated with Fasting blood sugar and insulin.
Lipid profile | Change from baseline cholesterol, triglyceride, high density lipoprotein, and low density lipoprotein at 12 weeks.
  Lipid profile will be measure by cholesterol, triglyceride, high density lipoprotein, and low density lipoprotein in mg/dl.
Tumor necrosis factor alpha, adiponectin, interleukin 1 beta, interleukin 6, brain derived neurotrophic factor, and malondialdehyde | Change from baseline tumor necrosis factor alpha, adiponectin, interleukin 1 beta, interleukin 6, brain derived neurotrophic factor, and malondialdehyde at 12 weeks.
  Tumor necrosis factor alpha, adiponectin, interleukin 1 beta, interleukin 6, brain derived neurotrophic factor, and malondialdehyde in pg/ml will be measure with ELISA assay kit.
Nitric oxide | Change from baseline Nitric oxide at 12 weeks.
  Nitric oxide in µM will measured with standard Griess reagents.

CONTACTS AND LOCATIONS:
Overall Officials: Daroonwan Suksom, Ph.D., Principal Investigator — Faculty of Sport Science Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided